CLINICAL TRIAL: NCT02222766
Title: Parents and Tots Together: A Family-Based Intervention to Promote Healthy Eating and Activity Behaviors Among Preschool Children
Brief Title: Parents and Tots Together: A Family-Based Obesity Prevention Intervention
Acronym: PTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: American Heart Association (Other); Harvard Medical School (HMS and HSDM) (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jess Haines, Associate Professor, University of Guelph
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 190331-41
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parents and Tots Together Program (Experimental): 9-week group-based parenting program
  Interventions: Behavioral: Parents and Tots Together Program
- Control (Active Comparator): Minimal attention control- weekly mailed information on general child development for 9 weeks
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Parents and Tots Together Program — Group-based parenting program, 9 sessions offered weekly
  Arms: Parents and Tots Together Program
Behavioral: Control — Minimal attention control- 9 weekly mailed information on general child development
  Arms: Control

SUMMARY:
The obesity epidemic has spared no age group, including our youngest children. My and others' formative research shows that ethnically-diverse, low-income parents of young children are enthusiastic about learning general parenting skills, such as discipline strategies, but less interested in nutrition and physical activity. To capitalize on this enthusiasm, I will create and test an intervention that embeds strategies to improve child weight-related behaviors within a general skills parenting program.

The overall goal of this study is to assess Parents and Tots Together (PTT), a family-based intervention to prevent obesity among children age 2 through 5 years. To achieve this goal, my colleagues and I will conduct a randomized controlled trial (RCT) among ethnically diverse, primarily low-income families. Our specific aims are to:

1. Determine the extent to which the intervention, compared with a control condition, results in a smaller age-associated increase in body mass index (BMI) among children after a 3- month intervention and a 9-month follow-up period (primary outcome).
2. Determine the extent to which the intervention, compared with a control condition, results in:

   1. Improved parent general parenting behaviors, i.e., increased use of positive discipline strategies.
   2. Improved parent feeding practices, i.e., increased responsiveness to child satiety cues.
   3. Improved child weight-related behaviors, i.e., increased sleep duration and physical activity, and reduced sugar-sweetened beverage intake and television/video viewing.

ELIGIBILITY:
Inclusion Criteria:

* parents who have a child aged 2-5 years
* respond to interviews and questionnaires in English or Spanish

Exclusion Criteria:

* any families who plan to move during the study period
* children or parents with severe health conditions that would prohibit them from participating in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI), adjusted for age and gender | baseline, post-intervention, 9-month follow-up

SECONDARY OUTCOMES:
Change in parent general parenting behaviors, i.e., use of positive discipline strategies. | baseline, post-intervention, 9-month follow-up
Change in child weight-related behaviors, i.e., sleep duration and physical activity, and sugar-sweetened beverage intake and television/video viewing. | baseline, post-intervention, 9-month follow-up
Change in parental feeding behaviors, i.e., controlling feeding practices | baseline, post-intervention, 9-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jess Haines, PhD, Principal Investigator — University of Guelph
Locations (1):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States